CLINICAL TRIAL: NCT06476379
Title: Can the Origin of Sperm - Ejaculated or Testicular- Affect Embryo Ploidy in Patients With Severe Male Factor Infertility?
Brief Title: Can the Origin of Sperm Affect Embryo Ploidy in Patients With Severe Male Factor Infertility?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFC-009
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-06

CONDITIONS: Male Infertility
Keywords: ICSI; Male infertility; PGT-A; TESE
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ejaculate (Active Comparator): Patients within this arm will undergo ICSI utilizing ejaculated sperm.
  Interventions: Other: Ejaculate
- Testicular (Active Comparator): Patients within this arm will undergo ICSI utilizing testicular sperm.
  Interventions: Procedure: Testicular sperm extraction (TESE)

INTERVENTIONS:
Procedure: Testicular sperm extraction (TESE) — Surgical procedure used to retrieve sperm directly from the testicles of men who have low sperm production or no sperm in their ejaculate
  Arms: Testicular
Other: Ejaculate — Ejaculate processing for ICSI
  Arms: Ejaculate

SUMMARY:
There is evidence indicating that sperm plays a role in determining blastocyst ploidy status. In our study, we aim to compare the outcomes of preimplantation genetic testing for aneuploidy (PGT-A) and the subsequent clinical outcomes following transfers of euploid embryos. This comparison will be conducted between cases where ejaculated sperm and cases where testicular sperm were used for intracytoplasmic sperm injection (ICSI), specifically focusing on severe male factor infertility patients.

ELIGIBILITY:
Inclusion Criteria:

* Cases planned to have ICSI PGT-A cycles
* Males diagnosed as severe male factor infertility
* Normo responder female partners

Exclusion Criteria:

* Leukocytospermia
* Presence of varicocele.
* Known genetic abnormality
* Use of sperm or oocyte donors
* Use of gestational carrier
* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Euploidy rate | 15 days post ICSI
  Defined as the proportion of euploid blastocysts
Aneuploidy rate | 15 days post ICSI
  Defined as the proportion of aneuploid blastocysts
Low mosaic rate | Time Frame: 15 days post ICSI
  Defined as the proportion of low mosaic blastocysts
High mosaic rate | Time Frame: 15 days post ICSI
  Defined as the proportion of high mosaic blastocysts
Implantation rate | 6-9 weeks post-embryo transfer
  defined as the percentage of successfully implanted embryos
Ongoing pregnancy rate | 12 weeks of gestation
  defined as a positive heartbeat on ultrasound beyond 12 weeks of gestation
Miscarriage rate | after 6 weeks of gestation
  defined as pregnancy loss following confirmation of clinical pregnancy
Clinical pregnancy rate | 6-9 weeks post-embryo transfer
  defined as the presence of a fetal heartbeat or gestational sac 6-9 weeks post-embryo transfer

SECONDARY OUTCOMES:
Fertilization rate | 1 day
  Defined as the proportion of fertilizaed oocytes
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3
Blastocyst development rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, Principal Investigator — Ganin Fertility Center; Hosam Zaki, FRCOG, Study Chair — Ganin Fertility Center; Refaat Gabre, PhD, Study Director — Faculty of Science, Cairo University; Mohamed Abbas, Study Chair — Cairo University; Nahla Osama, Phd, Study Chair — Faculty of Science, Cairo University
Locations (1):
- Ganin Fertility Center, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided